CLINICAL TRIAL: NCT02283658
Title: A Phase 2 Trial of Letrozole and Everolimus in Relapsed Hormone Receptor Positive Ovarian, Fallopian Tube or Primary Peritoneal Carcinomas
Brief Title: Everolimus and Letrozole in Treating Patients With Recurrent Hormone Receptor Positive Ovarian, Fallopian Tube, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1464; NCI-2014-02203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1464 (Other: Mayo Clinic in Florida); P30CA015083 (NIH)
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Ovarian Endometrioid Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Serous Surface Papillary Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Germ Cell Tumor; Recurrent Primary Peritoneal Carcinoma; Undifferentiated Ovarian Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Everolimus; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (everolimus and letrozole) (Experimental): Patients receive everolimus PO QD and letrozole PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Drug: Letrozole

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara

SUMMARY:
This pilot, phase II trial studies how well everolimus and letrozole work in treating patients with hormone receptor positive ovarian, fallopian tube, or primary peritoneal cavity cancer that has come back. Everolimus and letrozole may stop the growth of tumor cells by blocking some the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate that the combination of letrozole and everolimus leads to a higher percentage of patients who are free of progression at 12 weeks (PFS 12) as compared with that observed in a previously reported phase 2 trial of letrozole alone for relapsed ovarian carcinomas.

SECONDARY OBJECTIVES:

I. Cancer antigen (CA)-125 response, progression-free survival (PFS), overall survival (OS), the confirmed response rate, and adverse events.

TERTIARY OBJECTIVES:

I. Identify molecular biomarkers associated with a response to treatment with letrozole and everolimus in patients with relapsed ovarian carcinomas.

II. Develop and determine if response rates to letrozole and everolimus in patient derived xenograft (PDX) avatars correlate to responses noted in the patients.

OUTLINE:

Patients receive everolimus orally (PO) once daily (QD) and letrozole PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed estrogen receptor positive (greater than 10%) recurrent ovarian, fallopian tube or primary peritoneal carcinoma in post-menopausal women; note: pure clear cell and pure mucinous carcinomas are ineligible; both platinum sensitive, platinum resistant and platinum refractory disease are eligible; no limitations in the number of prior regimens
* Patient has disease amenable to biopsy and is agreeable to undergo a biopsy; note: under unusual circumstances, submission of ascites material may be acceptable if a biopsy is not possible; this will require approval by one of the study principal investigators
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 9.0 g/dL
* Total serum bilirubin =< 2 mg/dL
* Aspartate transaminase (AST) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN in patients with liver metastasis)
* International normalized ratio (INR) =< 2
* Creatinine =< 1.5 x ULN
* Fasting serum cholesterol =< 300 mg/dL or =< 7.75 mmol/L and fasting triglycerides =< 2.5 x ULN; in case of any of these thresholds be exceeded, the patient can only be included after initiation of appropriate lipid lowering medications
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide tissue samples for correlative research purposes

Exclusion Criteria:

* Any of the following

  * Pregnant women
  * Nursing women
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens including but not limited to any of the following that would limit compliance with study requirements:

  * Ongoing or active severe infection
  * Liver disease such as cirrhosis
  * Decompensated liver disease
  * Symptomatic congestive heart failure (New York heart Association class III or IV)
  * Unstable angina pectoris, serious uncontrolled cardiac arrhythmia, myocardial infarction =< 6 months prior to registration
  * Known severely impaired lung function (spirometry and diffusing capacity of the lung for carbon monoxide [DLCO] 50% or less of normal and oxygen [O2] saturation 88% or less at rest on room air)
  * Active bleeding diathesis
  * Psychiatric illness
* Known to be human immunodeficiency virus (HIV) positive
* Receiving any other investigational agent =< 4 weeks prior to registration which would be considered as treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; exceptions: non-melanotic skin cancer or carcinoma-in-situ of the cervix, uterus or breast; note: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* Patients currently receiving anticancer therapies or who have received anticancer therapies =< 4 weeks prior to registration (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral everolimus
* Uncontrolled diabetes mellitus as defined by hemoglobin (Hb)A1c > 8% despite adequate therapy; note: patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Chronic treatment with corticosteroids or other immunosuppressive agents; note: topical or inhaled corticosteroids are allowed
* Patients who have received live attenuated vaccines =< 1 week prior to registration and during the study; note: patient should also avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* History of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Prior therapy with everolimus or an aromatase inhibitor
* Known brain metastasis
* Active and chronic viral hepatitis (i.e. quantifiable serum hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B virus surface antigen [HBsAg], or quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA] in serum)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Colon-Otero, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Everolimus and Letrozole)
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One patient withdrew prior to treatment and was not included in any analysis.
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 60.0 [52.0 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive and Progression Free Survival at 12 Weeks
Description: The percentage of PFS12 successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated according to the exact binomial method. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), Disease progression in evaluable patients will be defined as one or more of the following:
  * Any new disease and/or clear progression of evaluable disease; OR
  * 2 fold elevation in CA-125 from its lowest level (either initial level or nadir, whichever is lowest, since study enrollment) combined with CA-125 elevation confirmed by re-assay at any time.
Time Frame: 12 weeks
Population: All evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
percentage of patients | 47 [24 to 71]

2. Secondary Outcome: Percentage of Participants With CA-125 Response
Description: CA-125 response: The key secondary endpoint of the study will be a CA-125 response, defined as a 50% or greater reduction in baseline CA-125. The null hypothesis will be set at CA-125 response rate of 8.3%, based on the response of single agent letrozole, as reported by Bowman et al (7). The treatment of letrozole and everolimus will be considered promising, based on CA-125, if the observed CA-125 response rate is 30% or more.
Time Frame: Up to 2 years
Population: All evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
percentage of patients | 21 [6 to 46]

3. Secondary Outcome: Confirmed Response Rate, Estimated Using RECIST 1.1 Criteria
Description: A confirmed tumor response is defined to be either a complete response or partial response noted as the objective status on 2 consecutive evaluations at least 4 weeks apart. A complete response (CR) in evaluable patients will be defined as:
  * Disappearance of any sign of (evaluable) disease, AND
  * Normalization of CA-125; if CA-125 normalizes, it should be confirmed at any time.
  A partial response (PR) in evaluable patients will be defined as:
  * Decrement in CA-125 by >50%, and
  * Improvement in any additional evaluable disease (if present) as assessed by the enrolling physician.
Time Frame: Up to 24 weeks
Population: All evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
percentage of patients | 16 [3 to 40]

4. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: The number of patients with adverse events.The maximum grade for each type of adverse event (AE) will be recorded for each patient, and frequency tables will be reviewed to determine AE patterns. These tables are reported in the adverse events section of this report.
Time Frame: Up to 30 days post-treatment
Population: All evaluable patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
Participants | 19

5. Secondary Outcome: Overall Suravival(OS)
Description: OS will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death from any cause, assessed up to 2 years
Population: All evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
Months | 13 [8.8 to NA] — Not Reached;Median was not reached due to too few PFS events.

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be estimated using the method of Kaplan-Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), Disease progression in evaluable patients will be defined as one or more of the following:
  Any new disease and/or clear progression of evaluable disease; OR 2 fold elevation in CA-125 from its lowest level (either initial level or nadir, whichever is lowest, since study enrollment) combined with CA-125 elevation confirmed by re-assay at any time.
Time Frame: Time from registration to the first of either disease progression or death from any cause, assessed up to 2 years
Population: All evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Everolimus and Letrozole)
Number analyzed (Participants) | 19
Months | 3.9 [2.8 to 11]

7. Other Pre Specified Outcome: Expression of Molecular Biomarkers Associated With a Response to Treatment With Letrozole and Everolimus in Patients With Relapsed Ovarian Carcinomas
Description: The Fisher's Exact test will be used to measure the associations.
Time Frame: 28 days following treatment initiation
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Response Rates to Letrozole and Everolimus in PDX Avatars
Description: Will determine if response rates to letrozole and everolimus in PDX avatars correlate to responses noted in the patients. The Fisher's Exact test will be used to measure the associations.
Time Frame: 28 days following treatment initiation
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Responsiveness of Tumors to Letrozole and Everolimus
Description: "Response" will be defined as tumors with at least a 50% reduction in tumor volume at study end. "Unresponsive" will be defined as tumors with less than 10% tumor volume reduction at study end. Intermediate values will be defined as "Stable". Tumor growth curves will be plotted graphically and notated to indicate the outcome status of the originating patients. End of study tumor volumes will be correlated with outcome status of the originating patient as well. The Fisher's Exact test will be used to measure the associations.
Time Frame: 28 days following treatment initiation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0.
Arm/Group | Treatment (Everolimus and Letrozole)
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Everolimus and Letrozole) (N=19)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Death NOS (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Everolimus and Letrozole) (N=19)
Anemia (Blood and lymphatic system disorders) | 7 (37)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Ascites (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 12 (28)
Esophageal ulcer (Gastrointestinal disorders) | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 14 (36)
Nausea (Gastrointestinal disorders) | 8 (17)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chills (General disorders) | 1 (13)
Edema limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 19 (89)
Fever (General disorders) | 1 (12)
Alanine aminotransferase increased (Investigations) | 2 (11)
Alkaline phosphatase increased (Investigations) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 4 (11)
Cholesterol high (Investigations) | 3 (23)
Neutrophil count decreased (Investigations) | 5 (14)
Platelet count decreased (Investigations) | 6 (28)
Urine output decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 4 (21)
Anorexia (Metabolism and nutrition disorders) | 6 (28)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (23)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3)
Dysgeusia (Nervous system disorders) | 1 (4)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (4)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (4)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (13)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (12)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes